CLINICAL TRIAL: NCT05389995
Title: Assessing the Effects of a Commercial Lemonade Beverage and Potassium Citrate on Urinary Stone Risk Factors
Brief Title: Potassium Citrate and Crystal Light Lemonade
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Amy Krambeck, Director of the Endourology/Stone Division, Northwestern University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: STU00216084
Record Dates: First submitted 2022-05-17; First posted 2022-05-25 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Kidney Stone
MeSH Terms: conditions — Kidney Calculi | interventions — Potassium Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Potassium citrate (Active Comparator)
  Interventions: Drug: Potassium citrate
- Crystal light (Active Comparator)
  Interventions: Drug: Crystal light
- Crystal light + potassium citrate (Active Comparator)
  Interventions: Drug: Potassium citrate + crystal light

INTERVENTIONS:
Drug: Potassium citrate — 7 days potassium citrate followed by 24 hour urine collection
  Arms: Potassium citrate
Drug: Crystal light — 7 days crystal light followed by 24 hour urine collection
  Arms: Crystal light
Drug: Potassium citrate + crystal light — 7 days potassium citrate + crystal light followed by 24 hour urine collection
  Arms: Crystal light + potassium citrate

SUMMARY:
To define the effect of crystal light, potassium citrate, or both on urinary stone risk factors in patients with a history of stone and hypocitraturia/low pH

ELIGIBILITY:
Inclusion Criteria:

1. Men and women between age 18-80 years
2. Willing to follow experimental protocol
3. Willing to complete 24-hour urine collections (three total)
4. Willing to sign the informed consent form
5. Completed Litholink Collection with blood work with results

   a. hypocitraturia OR aciduria i. Hypocitraturics must meet definition of < 450 mg/day for men < 550 mg/day for women.

   b. Low urine pH must be less than 5.6 c. potassium, BUN, creatinine, eGFR and hemoglobin A1c within normal limits

Exclusion Criteria:

1. Patients with severe hypocitraturia < 200 mg/day (men or women)
2. Patients with hyperkalemia, uncontrolled diabetes, chronic kidney disease, adrenal insufficiency, delayed gastric emptying (or drug induced delayed gastric emptying), peptic ulcer disease, or active UTI
3. Patients with distal renal tubular acidosis or medication induced RTA (e.g. carbonic anhydrase inhibitor, topiramate)
4. Members of vulnerable patient populations
5. Allergies to ingredients in crystal light
6. Patients lacking decisional capacity

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
urine citrate levels | Day 7 of week 1
  24 hour urine collection
urine citrate levels | Day 7 of week 3
  24 hour urine collection
urine citrate levels | Day 7 of week 5
  24 hour urine collection

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Chicago, Illinois, United States